CLINICAL TRIAL: NCT06885229
Title: Reuseable Face Masks to Reduce Risk of Viral Respiratory Infections and Exacerbations in Adults With Asthma: a Randomised Controlled Trial
Brief Title: Reusable Face Masks to Reduce Risk of Viral Respiratory Infections and Asthma Exacerbations
Acronym: REMASK
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Diminished minimum sample size needed to detect any effect of the intervention due to TwiCs study design, control arm participants were already recruited to the parent study (COVIDENCE UK).
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 176722; 352721 (Other: IRAS)
Record Dates: First submitted 2025-03-18; First posted 2025-03-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Infection; Asthma Exacerbations
Keywords: Upper Respiratory Infection; Acute Respiratory Infection; Asthma Exacerbation; Lower Respiratory Infection; Reusable Face Mask
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Offer of free reusable elastometic face mask and 12-month supply of replaceable filters to index participants with asthma and their adult household members
  Interventions: Device: FloMask - reuseable face mask
- Control (No Intervention): Usual asthma care without offer of intervention above

INTERVENTIONS:
Device: FloMask - reuseable face mask — Reuseable, elastomeric face mask with replaceable filters
  Arms: Intervention

SUMMARY:
REMASK trial is a Trial within Cohort study (TwiCs), nested within the COVIDENCE UK longitudinal study. It has been designed to determine whether the offer of a free reusable, elastomeric face mask to adults with asthma and other members of their household reduces risk of RT-PCR confirmed viral respiratory infections and asthma exacerbations.

ELIGIBILITY:
Eligibility criteria, participants with asthma ('index participants'):

Inclusion Criteria:

* Aged 16 or more years
* Doctor diagnosis of asthma
* Current prescription for treatment of asthma
* Participant in COVIDENCE UK nasal swab study

Exclusion Criteria:

* Regularly using any FFP-rated face mask when in an indoor public place
* Currently sharing household with one or more children
* Currently sharing household with one or more other COVIDENCE UK participants who have asthma
* Unable to tolerate wearing face mask

Eligibility criteria, household members of index participants:

Inclusion criteria

* Age 16 or more
* Living in same household as index participant who has consented to take part in trial

Exclusion criteria

- Unable to tolerate wearing face mask

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Time to first RT-PCR-proven viral respiratory infection | 12 months

SECONDARY OUTCOMES:
Time to first severe acute exacerbation of asthma (i.e. exacerbation requiring treatment with systemic corticosteroids and/or hospitalisation or emergency department visit) | 12 months
Time to first hospitalisation for treatment of acute respiratory infection or asthma exacerbation | 12 months
Time to first antibiotic prescription for treatment of acute respiratory infection | 12 months
Rate of RT-PCR-proven / symptom defined acute respiratory infections | 12 months
Cost per viral respiratory infection averted | 12 months
Cost per severe asthma exacerbation averted | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be shared with other researchers subject to terms of Data Transfer Agreement and IRB approval